CLINICAL TRIAL: NCT00118664
Title: Patient Plasma Response and Outcome in Septic Shock With Thrombocytopenia Associated Multiple Organ Failure in Children
Acronym: TAMOF
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 05-004
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Septic Shock; Thrombocytopenia; Multiple Organ Failure
Keywords: Septic Shock; Thrombocytopenia; Multiple Organ Failure; Pediatric
MeSH Terms: conditions — Shock, Septic; Thrombocytopenia; Multiple Organ Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to learn how blood clotting substances respond in children with septic shock, low platelet counts, and multiple organ failure (MOF) treated at different institutions.

Multiple organ failure can be related to an infection producing "septic shock," in which substances released in the blood cause poor blood flow to the organs. The number of platelets circulating in your child's blood stream is also decreased (this is called "thrombocytopenia") as a result of this condition. Research has shown that certain substances in the part of the blood known as plasma (the clear liquid part of the blood not including the red blood cells but holding blood clotting factors) can cause the organs to work poorly. The investigators would like to compare these blood responses in children with this condition, receiving a variety of different treatments, for multiple organ failure in other medical centers around the world. The investigators hope to enroll 80 patients into the study.

DETAILED DESCRIPTION:
Researchers have defined a subgroup of pediatric patients with critical illness who have a specific coagulation profile associated with thrombocytopenia. This distinct entity, defined as thrombocytopenia-associated multiple organ failure (TAMOF), has been demonstrated to predispose affected children to worsening organ failure and increased risk of death. A preliminary single-center study performed at Children's Hospital of Pittsburgh (CHP) suggested significant improvement in organ system dysfunction in TAMOF patients using a plasma exchange protocol compared to standard therapy alone. The investigators desire to further evaluate plasma profiles and clinical outcomes in pediatric TAMOF in a broader geographic setting. The investigators propose to perform a prospective multi-center observational cohort study to evaluate plasma response and clinical outcomes in pediatric patients with TAMOF due to critical illness associated with systemic infection, sepsis, organ transplant, chemotherapy or cardiopulmonary bypass. Plasma samples will be obtained from all patients for measurement of markers of coagulation and inflammation. The primary clinical endpoints measured will be organ failure index scores, pediatric logistic organ dysfunction (PELOD) scores, and days until resolution of organ failures. Cohort outcome analysis will also be performed by pairing patients at different centers receiving standard therapy with those receiving plasma exchange as an additional therapy.

ELIGIBILITY:
Inclusion Criteria:

All pediatric Intensive Care Unit (ICU) patients with the following inclusion criteria are eligible for enrollment:

* Weight > 5 kilograms (minimum weight required due to technical limits of exchange equipment)
* Multiple organ failure, defined as organ failure index (OFI) score > 3 present for < 30 hours
* Patients must have new (not present prior to admission) organ failure in at least 3 of the 5 organ systems.
* Thrombocytopenia (platelet count < 100,000 per ul), or in patients with a baseline platelet count < 100,000 per ul, a minimum 50% decrease in platelet count
* Etiology of MOF due to systemic infection, shock, transplantation, chemotherapy, or cardiopulmonary bypass

Exclusion Criteria:

* Treatment prior to study entry with any form of plasma exchange therapy within 30 days not for TAMOF
* Thrombocytopenia secondary to diagnosed thrombotic thrombocytopenic purpura/hemolytic uremic syndrome (TTP/HUS)
* Patients with terminal illness (i.e. not expected to live > 60 days even if they survive this acute illness) or in which withdrawal of therapy is being considered (do-not-resuscitate [DNR]/comfort measures only, limited therapy etc.)

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients admitted to a participating PICU.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2005-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D. Fortenberry, MD, Principal Investigator — Children's Healthcare of Atlanta
Locations (12):
- United States (12):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta at Egleston and Scottish Rite, Atlanta, Georgia
  - University of Iowa Children's Hospital, Iowa City, Iowa
  - LSU Health Sciences Center, Shreveport, Louisiana
  - University of Michigan Medical Center, Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Columbus Childrens Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Cook Children's Hospital, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No